CLINICAL TRIAL: NCT03513874
Title: The Effect of Metformin as add-on to Insulin in Non-obese Patients With Autoimmune Diabetes
Brief Title: Metformin Plus Insulin on Non-obese Autoimmune Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Director, Department of Endocrinology, Institute of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital, Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET201801
Record Dates: First submitted 2018-04-12; First posted 2018-05-02 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus; Autoimmune Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin + Insulin (Experimental)
  Interventions: Drug: Metformin; Drug: Insulin
- Insulin alone (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — Patients will be subscribed with 850mg metformin orally twice daily. Insulin will be continued as routine therapy.
  Arms: Metformin + Insulin
Drug: Insulin — Patients will continue insulin therapy following physicians' instructions.

SUMMARY:
The objective of this study is to evaluate the therapeutic effect of metformin as additional treatment with insulin on non-obese autoimmune diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to ADA criterias <5 years.
* Age≥ 18 years and less than 70 years.
* Non-obese: defined as BMI less than 28 kg/m2
* Positive for at least one of the anti-islet autoantibodies: GADA, IA2A, ZnT8A
* Fasting or postprandial plasma C-peptide more than 100 pmol/L
* Written informed consent from the patient or family representative.

Exclusion Criteria:

* History of any malignancy or other severe diseases
* Female patients who are pregnant or breastfeeding before or during the three-year follow-up
* Poor compliance or refusal to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean amplitude of glycemic excursions (MAGE) | 6 months
  MAGE is measured by applying continuous glucose monitoring system (CGMS) on subjects in each follow-up of this 6-month study.
Change in C-peptide | 6 months
  C-peptide are measured before and 2-hour after a mixed meal tolerance test at each follow-up of this study.

SECONDARY OUTCOMES:
Change in HbA1c | 6 months
Change in daily insulin dose | 6 months
Change in body mass index (BMI) | 6 months
Change in lipid profiles | 6 months
  Including triglyceride, total cholesterol, HDL-cholesterol and LDL-cholesterol
Adverse effects | 6 months
  Adverse effects are recorded at each time-point of the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China